CLINICAL TRIAL: NCT06893172
Title: Effectiveness of Warm Acupuncture for Postherpetic Neuralgia in the Context of the Qi Stagnation and Blood Stasis Syndrome: a Randomized Controlled Trial
Brief Title: Effectiveness of Warm Acupuncture in Patients with Postherpetic Neuralgia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Responsible Party: Principal Investigator, Dang Ngoc Ha Phuong, Investigator, University of Medicine and Pharmacy at Ho Chi Minh City
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1705/DHYD-HDDD
Record Dates: First submitted 2025-03-18; First posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Postherpetic Neuralgia ( PHN )
Keywords: Warm acupuncture; Postherpetic Neuralgia
MeSH Terms: conditions — Neuralgia, Postherpetic | interventions — Gabapentin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study Group (Experimental): The study group used gabapentin 300mg per tablet, twice a day, for a treatment period of 4 weeks, combined with Warm acupuncture at the Ashi point, EX-B2, LI4, TE6, PC5 and SP6, five times a week for 4 weeks.
  Interventions: Other: Warm acupuncture and Gabapentin
- Control Group (Active Comparator): The control group used gabapentin 300mg per tablet, twice a day, for a treatment period of 4 weeks
  Interventions: Drug: Gabapentin

INTERVENTIONS:
Other: Warm acupuncture and Gabapentin — This group used gabapentin 300mg per tablet, twice a day, for a treatment period of 4 weeks, combined with warm acupuncture at the Ashi point, EX-B2, LI4, TE6, PC5 and SP6, five times a week for 4 weeks.
  Arms: Study Group
Drug: Gabapentin — This group used gabapentin 300mg per tablet, twice a day, for a treatment period of 4 weeks
  Arms: Control Group

SUMMARY:
Postherpetic neuralgia (PHN) is the most common clinical complication of herpes zoster. PHN can persist for months to years, and in some cases, the pain may last for more than five years. Patients suffering from severe, prolonged pain endure significant distress, which seriously affects their quality of life and daily activities. Moreover, PHN can lead to insomnia, anxiety, depression, or even suicide. Currently, the treatment of PHN primarily focuses on pain management. First-line treatment options include gabapentin, pregabalin, tricyclic antidepressants, and 5% lidocaine patches.

Acupuncture is a widely used non-pharmacological therapy. A large number of clinical trials have demonstrated its effectiveness in treating various neuropathic pain conditions, including PHN. Acupuncture not only reduces pain perception but also alleviates anxiety and improves the quality of life for PHN patients. Among different acupuncture techniques, Warm Acupuncture (WA) is considered the most effective for treating peripheral neuropathic pain. Clinical case reports have also shown its pain-relieving effects in PHN patients.

However, there has been no study in Vietnam on the effectiveness of WA in pain reduction for patients with PHN. Therefore, this study is conducted to evaluate whether WA is effective in reducing pain and ensuring safety for treating PHN patients with Qi Stagnation and Blood Stasis syndrome. The findings will serve as a basis for the broader application of WA in the treatment of PHN.

DETAILED DESCRIPTION:
Patients with Postherpetic neuralgia in the trunk area, belonging to the Blood Stasis syndrome. They will be treated with a combination of Warm Acupuncture and Gabapentin.

The intervention period is four weeks. Warm Acupuncture will be performed five times a week and Gabapentin is administered daily for 4 weeks.

Data on the Visual Analog Scale (VAS), and side effects of Warm Acupuncture and Gabapentin will be recorded before the study and weekly for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with a history of herpes zoster in the trunk area.
* Individuals diagnosed with Postherpetic neuralgia (PHN) by a dermatologist, based on PHN diagnostic criteria, with pain persisting for 3 months or more after the skin lesions have healed.
* Individuals with a pain intensity score of ≥ 3, assessed using the Visual Analog Scale (VAS).
* Individuals diagnosed with Qi Stagnation and Blood Stasis syndrome by a Traditional Medicine doctor.
* Individuals aged 18 years or older.
* Individuals who volunteer to participate in the study and sign a consent form.

Exclusion Criteria:

* Active herpes zoster lesions, confirmed by the dermatologist treating the patient.
* Pregnant or breastfeeding women.
* Patients with severe cognitive impairment who cannot understand the study protocol.
* Patients with a history of allergy to Gabapentin.
* Currently participating in another interventional study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2025-08-29 (Estimated); Study Completion 2025-08-29 (Estimated)

PRIMARY OUTCOMES:
The change of the Visual Analog Scale (VAS) | Assessments were conducted before intervention and after each intervention week throughout the four weeks (Week 0, Week 1, Week 2, Week 3, Week 4)
  Pain will be measured using the Visual Analog Scale (VAS). Patients will be asked to circle a number from 0 to 10, where 0 represents "no pain" and 10 represents "the worst possible pain.

SECONDARY OUTCOMES:
Proportion of intervention-related adverse events | Up to four weeks
  While Warm acupuncture is generally considered safe, some patients may experience minor side effects at the application site. Studies on Warm Acupuncture have reported negligible adverse effects. The recorded adverse effects include burns, pain at the acupuncture site, and bleeding at the acupuncture site. The study will closely monitor and document any unexpected adverse events associated with the procedure.

REFERENCES:
- [Background] Zhao H, Nie W, Sun Y, Li S, Yang S, Meng F, Zhang L, Wang F, Huang S. Warm Needling Therapy and Acupuncture at Meridian-Sinew Sites Based on the Meridian-Sinew Theory: Hemiplegic Shoulder Pain. Evid Based Complement Alternat Med. 2015;2015:694973. doi: 10.1155/2015/694973. Epub 2015 Oct 1. PMID 26495023
- [Background] Li X, Han Y, Cui J, Yuan P, Di Z, Li L. Efficacy of Warm Needle Moxibustion on Lumbar Disc Herniation: A Meta-Analysis. J Evid Based Complementary Altern Med. 2016 Oct;21(4):311-9. doi: 10.1177/2156587215605419. Epub 2015 Sep 15. PMID 26378088
- [Background] Wang L, Qiu L, Zheng X, Ouyang J, Zhang M, He L, Zeng S, Liu B, Peng J. Effectiveness of electroacupuncture at Jiaji acupoints (EX-B2), plus moxibustion and intermediate on postherpetic neuralgia: a randomized controlled trial. J Tradit Chin Med. 2020 Feb;40(1):121-127. PMID 32227773
- [Background] Pei W, Zeng J, Lu L, Lin G, Ruan J. Is acupuncture an effective postherpetic neuralgia treatment? A systematic review and meta-analysis. J Pain Res. 2019 Jul 16;12:2155-2165. doi: 10.2147/JPR.S199950. eCollection 2019. PMID 31410050
- [Background] Zhao W, Huang H, Liu K, Wang S, Lin S, Long W, Li L, Zeng J, Lin G. Acupuncture and Moxibustion for Peripheral Neuropathic Pain: A Frequentist Network Meta-Analysis and Cost-Effectiveness Evaluation. Evid Based Complement Alternat Med. 2022 Mar 16;2022:6886465. doi: 10.1155/2022/6886465. eCollection 2022. PMID 35341147
- [Background] He K, Hu R, Huang Y, Qiu B, Chen Q, Ma R. Effects of Acupuncture on Neuropathic Pain Induced by Spinal Cord Injury: A Systematic Review and Meta-Analysis. Evid Based Complement Alternat Med. 2022 Aug 19;2022:6297484. doi: 10.1155/2022/6297484. eCollection 2022. PMID 36034938
- [Background] Johnson RW, Rice AS. Clinical practice. Postherpetic neuralgia. N Engl J Med. 2014 Oct 16;371(16):1526-33. doi: 10.1056/NEJMcp1403062. No abstract available. PMID 25317872
- [Background] Lin CS, Lin YC, Lao HC, Chen CC. Interventional Treatments for Postherpetic Neuralgia: A Systematic Review. Pain Physician. 2019 May;22(3):209-228. PMID 31151330
- [Background] Zhang M, Gao CX, Ma KT, Li L, Dai ZG, Wang S, Si JQ. A Meta-Analysis of Therapeutic Efficacy and Safety of Gabapentin in the Treatment of Postherpetic Neuralgia from Randomized Controlled Trials. Biomed Res Int. 2018 Jul 4;2018:7474207. doi: 10.1155/2018/7474207. eCollection 2018. PMID 30069477
- [Background] Du J, Sun G, Ma H, Xiang P, Guo Y, Deng Y, Li S, Li X. Prevalence and Risk Factors of Anxiety and Depression in Patients with Postherpetic Neuralgia: A Retrospective Study. Dermatology. 2021;237(6):891-895. doi: 10.1159/000512190. Epub 2020 Dec 16. PMID 33326962
- [Background] Putri Mellaratna W, Jusuf NK, Yosi A. The impact of pain intensity on quality of life of postherpetic neuralgia patients. Med Glas (Zenica). 2020 Aug 1;17(2):439-444. doi: 10.17392/1111-20. PMID 32253903
- [Background] Yang F, Yu S, Fan B, Liu Y, Chen YX, Kudel I, Concialdi K, DiBonaventura M, Hopps M, Hlavacek P, Cappelleri JC, Sadosky A, Parsons B, Udall M. The Epidemiology of Herpes Zoster and Postherpetic Neuralgia in China: Results from a Cross-Sectional Study. Pain Ther. 2019 Dec;8(2):249-259. doi: 10.1007/s40122-019-0127-z. Epub 2019 Jun 19. PMID 31218562
- [Background] Harpaz R, Ortega-Sanchez IR, Seward JF; Advisory Committee on Immunization Practices (ACIP) Centers for Disease Control and Prevention (CDC). Prevention of herpes zoster: recommendations of the Advisory Committee on Immunization Practices (ACIP). MMWR Recomm Rep. 2008 Jun 6;57(RR-5):1-30; quiz CE2-4. PMID 18528318
- [Background] Lin YH, Huang LM, Chang IS, Tsai FY, Lu CY, Shao PL, Chang LY; Varicella-Zoster Working Group; Advisory Committee on Immunization Practices, Taiwan. Disease burden and epidemiology of herpes zoster in pre-vaccine Taiwan. Vaccine. 2010 Feb 3;28(5):1217-20. doi: 10.1016/j.vaccine.2009.11.029. Epub 2009 Nov 26. PMID 19944790
- [Background] Chen LK, Arai H, Chen LY, Chou MY, Djauzi S, Dong B, Kojima T, Kwon KT, Leong HN, Leung EM, Liang CK, Liu X, Mathai D, Pan JY, Peng LN, Poblete ER, Poi PJ, Reid S, Tantawichien T, Won CW. Looking back to move forward: a twenty-year audit of herpes zoster in Asia-Pacific. BMC Infect Dis. 2017 Mar 15;17(1):213. doi: 10.1186/s12879-017-2198-y. PMID 28298208